CLINICAL TRIAL: NCT02731651
Title: Effect of CO2 Pneumoperitoneum on Human Ovary: Preliminary Study
Brief Title: Effect of Pneumoperitoneum on Human Ovary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ali Akdemir, MD, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AAkdemir2
Record Dates: First submitted 2016-03-23; First posted 2016-04-07 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Open Hysterectomy (Active Comparator): Open hysterectomy was performed with taking one of the ovaries at the beginning and the other ovary was removed at the end of the surgery.
  Interventions: Procedure: open hysterectomy
- LaparoscopicAssistedVaginalHysterectomy (Active Comparator): Surgery in Group 2 (LAVH): Laparoscopic Assisted Vaginal Hysterectomy was performed with taking one of the ovary at the beginning of the procedure and the other ovary was removed at the end of the surgery.
  Interventions: Procedure: laparoscopic assisted vaginal hysterectomy

INTERVENTIONS:
Procedure: open hysterectomy — Hysterectomy with laparotomy incision.
  Arms: Open Hysterectomy
Procedure: laparoscopic assisted vaginal hysterectomy — Hysterectomy with laparoscopic assisstance.
  Arms: LaparoscopicAssistedVaginalHysterectomy

SUMMARY:
Laparoscopic surgery has played a pivotal role in all surgical fields in modern medicine. It has some well known advantages over open surgery. For this reason laparoscopic surgery is know the first choice for many surgical procedures, even in gynecology. On the other hand, despite the advantages of laparoscopy carbon dioxide (CO2) pneumoperitoneum is not free from side effects. Experimental studies and limited clinical studies showed that pneumoperitoneum leads to a decrease in the blood flow to intra-abdominal organs during laparoscopic surgery. This is also known as ischemia, leads to the production of free O2 radicals. The desufflation of the abdominal cavity at the end of the procedure reduces the increased abdominal pressure and increase the perfusion of intra-abdominal organs. However this will not stop the production of free radicals. This reperfusion period even exaggerate the release of free radicals. This phenomenon is called as ischemia/reperfusion (I/R) model that leads to release of various free radicals, which are the most important mediators of oxidative tissue injury and consequential organ dysfunction. Recently both oxidative tissue injury and consequential dysfunction have been shown in ovarian tissue in experimental animal studies. But the data related to human ovary is still scarce. Thus the aim of the study is to evaluate the effect of I/R injury related to CO2 pneumoperitoneum on human ovary.

DETAILED DESCRIPTION:
Twenty patients at premenopausal period and with an indication of hysterectomy with benign uterine pathology were included in the study.

Patients were randomly assigned to open hysterectomy (group 1) and laparoscopic assisted vaginal hysterectomy (group 2).

In all patients, surgeries were performed under endotracheal general anesthesia with mechanical ventilation. Under the general anesthesia Arterial blood gas, airway pressure, dynamic pulmonary compliance, peripheral pulse-oximetry, end tidal carbon dioxide pressure level (set at between 35 and 45 mm/hg), blood pressure, and cardiac rhythm were monitored continuously during the surgery. All patients received a single dose of cefazolin sodium as a prophylactic antibiotic. Low molecular weight heparin was not given the patients.

Surgery in Group 1 (open hysterectomy) After the induction of the anesthesia and before the skin incision first venous blood sample was collected. Abdominal access was performed with Pfannenstiel incision. One of the ovaries was excised at the initial step. Contralateral utero-ovarian ligament and bilateral round ligaments were then ligated and transected. After the identification of the anterior and posterior leaves of the broad ligament, bladder flap was developed and bladder was moved off the lower uterine segment. Bilateral vascular uterine pedicles, and sacro uterine ligaments were ligated and transected. After performing circumferential colpotomy vaginal cuff was closed. At the final step, before closing the abdominal incision contralateral ovary was excised. Both ovaries were macroscopically evaluated by an expert pathologist immediately after their excision. Before the preparation of the ovaries for histopathological evaluation, 1 cm3 piece of each ovary was excised for biochemical evaluation of the malondialdehyde (MDA) level. Second blood sample was collected immediately after the skin closure.

Surgery in Group 2 (LAVH) After the induction of the general anesthesia and before skin incision first venous blood sample was collected from the patients. This blood sample was reflected the baseline status. After umbilical skin incision was made, pneumoperitoneum was created via veress needle using a nonheated (room temperature) and dry CO2. A 10 mm trocar was then inserted into the abdominal cavity through umbilical incision for optic system. Three 5 mm ancillary trocars were then inserted under direct vision. Two were in lower abdominal quadrants and one on the left side of the umbilicus. Intraabdominal pressure (IAP) pressure was set at 14 mmHg and maintained. Immediately after the port placement one of the ovaries was excised in a few minutes. Surgery was continued with ligating and transecting contralateral utero-ovarian ligament and bilateral round ligaments. (Contralateral infundibulopelvic ligament (IP), which contains the main vascular supply of the ovary, was not ligated and transected at this step, ligating and transecting of the IP was performed at the end of the procedure.) Anterior and posterior leaves of the broad ligaments were then identified and bladder flap was developed and the bladder was mobilized off the lower uterine segment. At this point pneumoperitoneum was released and the surgical team performed the rest of the procedure vaginally. Before releasing the pneumoperitoneum second blood sample was collected to reflecting the ischemic status. Circumferential colpotomy was performed and bilateral sacro-uterine ligaments and uterine vascular pedicles were ligated and transected vaginally. Vaginal cuff was closed vaginally. At this point pneumoperitoneum was achieved again to excise the contralateral ovary in a few minutes. Before pneumoperitoneum was performed again third blood sample was collected to represent the reperfusion status. Both ovaries were macroscopically evaluated by an expert pathologist immediately after their excision. Before the preparation of the ovaries for histopathological evaluation, 1 cm3 piece of each ovary was excised for biochemical evaluation of the malondialdehyde (MDA) level. In this group, the first excised ovary represented the baseline status, and the other ovary (excised at the end of the procedure) was exposed to the ischemia and reperfusion condition and represented the I/R status.

Plasma MDA and 8-hydroxy-2' -deoxyguanosine (8OHdG) was measured as a marker of oxidative stress. Ovarian tissue MDA level was also measured as a marker of tissue oxidative stress. Besides, ovarian histopathological examination was performed to score the oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* patients with an indication of hysterectomy with benign uterine pathology

Exclusion Criteria:

* patients with cardio vascular, pulmonary , hepatic or renal dysfunction,
* previous abdominal surgery,
* morbid obesity,
* intraabdominal adhesions preventing removal of the first ovary in a few minutes,
* any ovarian disease,
* current smoker, and
* refusal to participation.

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Evaluating the ischemia reperfusion injury related to pneumoperitoneum on human ovary. | 1 day
  Ischemia reperfusion injury was evaluated with histopathological assessment, and with assessing ovarian tissue malondialdehyde levels biochemically.

IPD SHARING:
Plan to Share IPD: Undecided